CLINICAL TRIAL: NCT04302207
Title: The ROUTT-B (Reduce Over-Utilized Tests and Treatments in Bronchiolitis) Study: Developing a Roadmap for De-Implementation
Brief Title: The ROUTT-B (Reduce Over-Utilized Tests and Treatments in Bronchiolitis) Study
Acronym: ROUTT-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19-0728
Record Dates: First submitted 2020-02-19; First posted 2020-03-10 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Intervention Model Description: non-randomized controlled trial of ROUTT-B using a parallel experimental and control interrupted time series study design extending over baseline, intervention, and post-intervention period.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High use hospitals (Experimental): patients 1-23 months with Bronchiolitis seen in emergency department, urgent care or admitted patients will be included; provider surveys measuring the acceptability, appropriateness, feasibility, and perceived burden of piloted strategies; review of patient data extracted from electronic health record to include baseline, intervention and post-intervention data
  Interventions: Behavioral: De-implementation Strategy for Bronchiolitis
- Low use hospital (Children's Hospital Colorado) (No Intervention): patients 1-23 months with Bronchiolitis seen in emergency department, urgent care or admitted patients will be included; review of patient data extracted from electronic health record to include data over the same time periods as the experimental groups' baseline, intervention, and post-intervention data

INTERVENTIONS:
Behavioral: De-implementation Strategy for Bronchiolitis — De-implementation strategy to reduce over-use of treatments for patients with bronchiolitis
  Arms: High use hospitals

SUMMARY:
Over-testing and over-treatment costs the US healthcare system hundreds of billions of dollars a year, and has measurable negative impacts on patients' physical, emotional, and financial health making it a significant public health concern. The proposed research will advance "de-implementation" science by identifying processes and strategies to stop or reduce over-testing and over-treatment that can be broadly adapted to varied contexts and disease processes to improve the delivery of guideline concordant, evidence-based care and improve patient outcomes.

DETAILED DESCRIPTION:
The overarching goal of this proposal is to use bronchiolitis as a case study to advance the science of de-implementation by identifying strategies and processes for reducing over-testing and over-treatment in bronchiolitis that can later be broadly adapted to varied contexts and disease processes. The challenge in bronchiolitis is that providing high-quality, evidenced-based care requires a "less is more" approach as the non- recommended, outdated, and potentially harmful tests and treatments that most admitted patients receive do not have replacements. Therefore, bronchiolitis which is the most common cause of hospitalization among infants, is an ideal condition to study de-implementation.

In her set of projects, Dr. Tyler proposes the innovative application of dissemination and implementation (D&I) science to the unique problem of de-implementation. Within a learning health system called PEDSnet, Dr. Tyler will use the PRISM D&I model as a guide to: 1) use qualitative methods to define contextual factors influencing over-utilization in bronchiolitis from the perspective of healthcare providers, parents, and healthcare organizations, 2) develop a set of pragmatic, feasible, and effective de-implementation strategies for bronchiolitis that includes guidance on how to adapt the strategies to local contexts, and 3) conduct a pilot study to determine the feasibility, acceptability, and de-implementation effectiveness of the de-implementation strategies. As one of the first explorations of contextual factors fostering overuse or enabling successful de-implementation, this study is expected to generate valuable knowledge relevant to de- implementation across diseases and healthcare settings. The results will provide pilot data for a large-scale, pragmatic, randomized-controlled trial of the de-implementation strategies so that ineffective and potentially harmful medical practices are reduced.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 1-23 months seen at a participating site for bronchiolitis
* Providers at participating sites that see eligible patients (defined above)
* Parents who have an eligible child at participating study sites (parent interviews)

Exclusion Criteria:

* Patients outside the age limits and do not have bronchiolitis
* Providers not at participating site
* Parents who do not have an eligible child at participating study site.

Ages: 1 Month to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Using survey instruments developed by the research team, measure acceptability of the de-implementation strategies for bronchiolitis patients at high-use hospital | through study completion, an average of 1 year
  Online surveys will be given to providers care team members that experience the de-implementation strategies at the high-use hospitals to determine acceptability and appropriateness

SECONDARY OUTCOMES:
Measure de-implementation effectiveness | through study completion, an average of 1 year
  Looking at electronic health records, review the change in the utilization rates of CXR, bronchodilators, and VT for patients affected with bronchiolitis at all hospitals
Measure feasibility of deploying ROUTT-B from the perspectives of the quality improvement team who will deploy it. | through study completion, an average of 1 year
  Measured through mixed methods approach (qualitative interviews or focus groups and provider surveys)

OTHER OUTCOMES:
Proportion of patients receiving antibiotics | through study completion, an average of 1 year
  using electronic health records of patient population at both hospitals
Median length of hospitalization in hours | through study completion, an average of 1 year
  using electronic health records of patient population at all hospitals
Unintended consequences | through study completion, an average of 1 year
  7 day ED/UC all cause revisits, 7 day all cause readmissions, ICU level care at index visit at all hospitals
Stakeholders' perceptions of impact on patient outcomes | through study completion, an average of 1 year
  measured through provider and care team survey at high-use hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tyler, MD, Principal Investigator — Nationwide Children's Hospital
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - Nationwide Children's Hospital, Columbus, Ohio
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tyler A, Krack P, Bakel LA, O'Hara K, Scudamore D, Topoz I, Freeman J, Moss A, Allen R, Swanson A, Bajaj L. Interventions to Reduce Over-Utilized Tests and Treatments in Bronchiolitis. Pediatrics. 2018 Jun;141(6):e20170485. doi: 10.1542/peds.2017-0485. Epub 2018 May 11. PMID 29752289